CLINICAL TRIAL: NCT06839859
Title: An Online Family-based Program to Reduce Inequity Among Sexual and Gender Minority Youth of Color (Pilot RCT)
Brief Title: Family Acceptance Project Online (Pilot RCT)
Acronym: FAP-O
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Nebraska Lincoln (Other); University of Colorado, Colorado Springs (Other)
Responsible Party: Principal Investigator, Katie M Edwards, Professor, School of Social Work, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00264028; 203677 (Other Grant/Funding Number: William T Grant Foundation)
Record Dates: First submitted 2025-02-07; First posted 2025-02-21 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: LGBTQ; Racial Disparities; Family Relationships; Minority Stress; Depression; Anxiety; Drug Use; Teen Dating Violence; Sexual Risk Reduction
Keywords: LGBTQ; Family Support; Parents of LGBTQ Youth; Racial/Ethnic Minority; Health Equity; Family Acceptance
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study involves n=90 dyads (caregiver/LGBTQ+ youth) randomly assigned to treatment group or wait-list control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Experimental): Participants in this arm receive the intervention (9, 2-hour weekly sessions) immediately after enrollment
  Interventions: Behavioral: Family Acceptance Project - Online
- Waitlist Control (No Intervention): Provide check-ins, provide resources, and offer participants in this arm the same intervention program as the experimental immediate treatment group after 6-month follow-ups and measurements have been completed.

INTERVENTIONS:
Behavioral: Family Acceptance Project - Online — a 9-week long online group program for LGBTQ+ youth of color and their parents / caregivers
  Arms: Immediate Treatment

SUMMARY:
Research shows that sexual and gender minority youth (SGMY) experience high rates of mental health problems and other challenges (e.g., social, academic). A major factor that leads to these challenges is family rejection (family behaviors and reactions that minimize, deny, ridicule and attempt to prevent or change a child's sexual orientation, gender identity and gender expression). Racial and ethnic minority youth experience the highest rates of family rejection and related health risks.

The Family Acceptance Project (FAP) is a research, education, and intervention initiative that was founded more than 20 years ago to help diverse families learn to support and affirm their SGMY. FAP's Family Support Model is grounded in the lived experiences of diverse SGMY and families and uses a culture-based family support framework that enables parents and caregivers to change rejecting behaviors that FAP's research has shown contribute to health risks and increase supportive and accepting behaviors that promote well-being for SGMY.

The overall goal of this research project is to evaluate a nine-week online version of FAP's Family Support Model (FAP-O). The investigators will specifically study how FAP-O:

1. Promotes parent/caregiver acceptance and support of their sexual and gender minority youth.
2. Increases family bonding and communication.
3. Increases SGMYs' feelings of pride in being LGBTQ+ and more hopeful about the future.
4. Leads to reductions in mental health problems reported by SGMY who experience family rejection.

Before receiving FAP-O's family support services, racial and ethnic minority SGMY (ages 14 to 25) and their caregivers will complete an initial pre-test survey. After completing this initial (baseline) survey, half of the families will participate in program sessions. Following the first round of sessions, all participants will complete an immediate follow-up survey, with an additional survey conducted six months after this. These surveys help us learn if FAP-O impacts the project's goals above. After the final survey, the other half of the families will attend program sessions. The investigators will also ask SGMY and caregivers to share what they liked about the program and their guidance for enhancing it.

DETAILED DESCRIPTION:
Research documents epidemic rates of behavioral (e.g., alcohol use), emotional (e.g., depression, suicidality), relational (e.g., dating violence victimization and perpetration), and academic (e.g., academic commitment) problems among sexual and gender minority youth (SGMY), including SGMY of color who experience disproportionate inequities due to their multiply minoritized status.

The disproportionally high rates of behavioral, emotional, relational, and academic problems among SGMY can be explained by experiences of minority stress related to oppression and discrimination specific to occupying minoritized social identities, including sexual orientation, gender identity, and race/ethnicity. Research shows that racial discrimination, SOGIE (sexual orientation, gender identity, and expression) discrimination and victimization interact to exacerbate their negative associations on deleterious behavioral, emotional, relational, and academic outcomes.

Families, including caregivers, play a critical role in the lives of SGMY by buffering against, exacerbating, and/or serving as a direct source of minority stress. A prevalent form of minority stress experienced by SGMY is family rejection (attitudes and behaviors that demonstrate disapproval of and/or efforts to change one's child's SOGIE) related to their sexual/gender minority identity. Indeed, 71% to 82% of SGMY report family rejection, and family rejection is more pronounced among SGMY of color (compared to white, non-Latinx SGMY).

Family rejection predicts a host of deleterious emotional, behavioral, relational, and academic outcomes. For example, youth who are told by their caregivers that something is inherently wrong with them, that they will never have a good future, and engage in damaging behaviors (e.g., expulsion from the home, harsh parenting/abuse), may internalize those experiences. This internalization may result in depression and suicidality. Caregiver rejection may also lead to risk behaviors in SGMY via the lack of positive parent-child relationships, poor communication, absence of modeling of healthy attitudes and behaviors, and poor monitoring/supervision. The absence of these parenting behaviors and parent-child relationship variables may lead to substance use (via poor coping mechanisms and/or lack of parental monitoring) as well as sexual risk taking and/or dating violence (via lack of knowledge about healthy relationship behaviors, the inability to seek guidance about mistreatment from others, and due to internalized oppression which may render SGMY more vulnerable to victimization and less likely to leave an abusive relationship).

The etiology of caregiver rejection of their SGMY is complex and multifaceted, Caregivers may engage in rejecting behaviors due to care for their SGMY and desire to help their child "fit in", "have a good life", and "be accepted by others" as well as a lack of information on SOGIE and/or how to support their SGMY. Caregiver rejection of their SGMY is often rooted in negative societal, cultural, and/or religious views about SGM people, including strict notions about gender.

Beyond caregiver acceptance (a key component of reducing inequality among SGMY and promoting positive youth development [PYD]), SGMY of color who report a strong sense of connection to other SGM individuals have better outcomes than SGMY of color who do not report these connections. Thus, programs that simultaneously seek to reduce caregiver rejection of their SGMY and provide opportunities for SGMY to connect with other SGMY may be especially powerful in reducing minority stressors and deleterious outcomes and promoting overall PYD. What is more, programs that provide accurate information about SOGIE, teach caregivers how to advocate for their SGMY, and reduce internalized oppression among SGMY may also foster the development of critical consciousness (i.e., the process of understanding social conditions, health inequities, and systems of oppression) in SGMY of color and their caregivers. Critical consciousness not only fosters thriving in the face of adversity but also may lead to action (e.g., vocalizing the need for policy change) to reduce inequality.

The Family Acceptance Project

The Family Acceptance Project (FAP) is a rigorously developed family-based intervention for caregivers of SGMY as well as SGMY (within the context of their families) in the U.S. FAP seeks to prevent myriad deleterious outcomes and promote PYD for SGMY in the context of their families, cultures, and faith communities. FAP is designed to help families via caregivers to decrease rejection and to support and affirm their SGMY (thereby reducing SGMY behavioral, social, emotional, relational, and academic problems). Whereas to date FAP has been almost exclusively delivered in in-person formats, a highly innovative component of the current project is to create an online version of FAP.

FAP includes both caregiver and SGMY components as well as family and group sessions. Work with caregivers focuses on 1) assessing caregivers' reactions to their SGMY; 2) providing psychoeducation about family accepting and rejecting behaviors in the context of their cultural and religious values; and 3) teaching skills to show love and affirmation and acceptance to ones' SGMY as well as advocacy skills to stand up for their SGMY in the face rejection. Youth components focus on 1) psychoeducation on family rejecting and accepting behaviors, 2) reducing internalized oppression and increasing positive identity development, and 3) instilling hope for the future. FAP also offers opportunities to build connections with others (e.g., caregiver peer support, LGBTQ+ sense of community among SGMY) and promotes family bonding and communication, all of which is hypothesized to reduce internalized oppression among SGMY and promote their PYD.

In FAP, education and guidance are presented to program participants in ways that resonate with caregivers' cultural and religious values. This allows caregivers to decrease rejecting behaviors that increase risk and increase supportive behaviors that help to protect against risk and support well-being. FAP helps caregivers to develop a different way of thinking about their SGMY that moves from issues of morality to those focused on ensuring the health and well-being of their SGMY. FAP helps youth to understand how their family's cultural and religious beliefs impact their sense of self-worth, their risk behaviors, and hope for the future. Many SGMY see family rejecting behaviors as the price of staying connected to their family, their culture, and their faith. In addition to learning about chosen family, learning that caregivers can change their behavior and learn to support and accept them is liberating and motivates youth to deepen family connections and invest in these relationships.

Despite its national recognition and reach, there is little research evaluating the efficacy of FAP. There is an urgent need for rigorous research on FAP to document its efficacy in reducing behavioral, social, emotional, relational, and academic problems especially among SGMY of color for whom FAP was largely developed. Moreover, FAP was initially developed for in-person delivery. Yet, there is also a need for research that examines innovative methods (e.g., online delivery) for implementation so that FAP can reach SGMY of color across the U.S., including rural regions of the U.S. where access to affirming, family-based interventions to support SGMY are rare if nonexistent.

The aim of the current study is to evaluate FAP-O via a randomized control trial (RCT) of caregiver-SGMY of color (ages 14 to 25) dyads (45 dyads assigned to the FAP-O and 45 dyads assigned to the waitlist control condition), assess the acceptability and feasibility of the FAP-O via program observations, post-session surveys (n = 90 dyads), and exit interviews (n=20) with SGMY of color and their caregiver(s). Test the FAP-O's efficacy in reducing behavioral, emotional, relational, and academic problems via a baseline survey followed by an immediate post-test and 6-month follow-up survey. Identify mediators (e.g., increases in family bonding, reductions in internalized oppression, decreases in rejection and increases in acceptance of SGMY by caregivers, increases in positive ethnic/racial identities) and examine intervention promise among demographic subgroups (e.g., race and ethnicity, gender identity, sexual identity, religiosity) and those experiencing low or high levels of racial or ethnic discrimination via surveys.

ELIGIBILITY:
Inclusion Criteria (youth):

1. Identify as a sexual/gender minority (including youth questioning their sexual orientation and/or gender identity AND their identity must be known to their participating caregiver).
2. Identify as a person of color/belonging to a minority racial and/or ethnic group.
3. Be between the ages of 14 and 25 years
4. Read and speak English
5. Live in the United States
6. Report consistent access to a phone, tablet, and/or computer with high-speed internet access
7. Report an ability to attend eight, two-hour online sessions at pre-determined times
8. Report moderate to high levels of caregiver/family rejection
9. Not be at high-risk for suicide
10. Not be actively psychotic

Inclusion Criteria (caregivers):

1. Be a caregiver (biological parent, stepparent, grandparent, aunt/uncle, or another adult who provides care) to an SGMY of color between the ages of 14 to 25
2. Be over the age of 18
3. Read and speak English
4. Live in the United States
5. Report consistent access to a phone, tablet, and/or computer with high-speed internet access.
6. Report an ability to attend nine, two-hour online sessions at pre-determined times.
7. Be aware of the SGM youth's minority identity
8. NOT identify as SGM
9. Report spending time with participating youth at least 5 waking hours per week
10. Not be at high-risk for suicide
11. Not be actively psychotic

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Depression (Youth and Caregivers) | Past 2-weeks at pre-test (enrollment), past 2-weeks at post-test (within one week of intervention end), past 2-weeks at 6-month follow-up
  Patient Health Questionnaire (PHQ-9) modified- 9 Item measure for detecting major depression. Measured on a 4 point scale with 0= Not at all to 3= Nearly every day. Higher scores indicate more depressive symptomology.
Suicidality (Youth) | Past month at pre-test (enrollment), past month at post-test (within one week of intervention end), past month at 6-month follow-up
  The Suicidal Ideation Attributes Scale (SIDAS): Community-based validation study of a new scale for the measurement of suicidal ideation. Suicide and Life-Threatening Behavior. A 5 item measure. Scale is 0-10 with higher scores indicating severity of suicidal ideation.
Generalized Anxiety (Youth and Caregivers) | Past 2-weeks at pre-test (enrollment), past 2-weeks at post-test (within one week of intervention end), past 2-weeks at 6-month follow-up
  Generalized Anxiety Disorder Screener (GAD-7) is a self-report anxiety questionnaire of 7 items. The 4 point scale is 0= Not at all to 3= Nearly every day. Higher scores signify greater anxiety severity.
Alcohol Use (Youth) | Past month at pre-test (enrollment), past month at post-test (within one week of intervention end), past month at 6-month follow-up
  Youth Risk Behavior Survey 2023 - Alcohol items is a 3 item measure that assesses alcohol use over the past 30 days. item 1 is a 7 point scale 0=0 days to 6= all 30 days, item 2 is a 7 point scale 0=0 days to 6= 20 or more days, and item 3 is an 8 point scale 0=I did not drink alcohol in the past 30 days to 7=10 or more drinks. Higher scores represent more alcohol use.
Drug Use (Youth) | Past month at pre-test (enrollment), past month at post-test (within one week of intervention end), past month at 6-month follow-up
  Youth Risk Behavior Survey 2023 - Drug use items is an 8 item measure of drug use over the past 30 days. The 6 point scale 0=0 times to 5=40 or more times. Higher scores represent more drug use.
Teen Dating Violence - Victimization (Youth) | Past month at pre-test (enrollment), past month at post-test (within one week of intervention end), past month at 6-month follow-up
  Measure of Adolescent Relationship Harassment and Abuse (MARSHA) - Victimization a 21 item measure with 3 subscales (privacy, social, intimidation) a 4 point scale with 0= 0 times to 3= more than 10 times. Higher scores indicate presence of unhealthy relationship behavior victimization.
Teen Dating Violence - Perpetration (Youth) | Past month at pre-test (enrollment), past month at post-test (within one week of intervention end), past month at 6-month follow-up
  Measure of Adolescent Relationship Harassment and Abuse (MARSHA) - Perpetration 24 item measure with 4 subscales (social, intimidation, cyber control, isolation). 4 point scale with 0= 0 times to 3= more than 10 times. Higher scores indicate unhealthy relationship behavior perpetration.
School Engagement (Youth) | No time frame at pre-test (enrollment), post-test (within one week of intervention end), or 6-month follow-up.
  Items from Hulsey et al. (2018) is a 5 item measure with a 4 point scale 1=Not at all true of me -- 4= Extremely true of me. Higher scores indicate increased school engagement.
Sexual Risk Taking (Youth) | Past month at pre-test (enrollment), past month at post-test (within one week of intervention end), past month at 6-month follow-up
  Youth Risk Behavior Survey 2023 - Sexual risk taking items over the past 30 days is a 4 item measure with item 1 having an 11 point scale 0= I have never had sex/I have had sex, but not in the past month to 10= 10 or more people and the remaining 3 items have a 5 point scale 0= 0 times to 4= 6 or more times. Higher scores indicate higher risky sexual behavior.
Caregiver perspective of youth mental health (Caregivers) | No time frame at pre-test (enrollment), post-test (withing one week of intervention end), or 6-month follow-up.
  Pediatric Symptom Checklist-17 (PSC-17) is a 17 item measure with a 3 point scale 0=Never to 2=Often. Higher scores can indicate mental health disorder characteristics.

OTHER OUTCOMES:
(Intermediary Outcome) Caregiver Accepting and Rejecting Behaviors (Youth and Caregivers) | Time Frame: Past month at pre-test (enrollment), past month at post-test (within one week of intervention end), past month at 6-month follow-up
  FAP-Reactions, Advocacy, Feelings/Experiences is a 34 item measure with a 4 point scale for items 1-30 0=Never to 3=Many times. Higher scores indicate more accepting behavior. A 5 point scale for items 31-32 1=Very Upset to 5=Very Happy with higher scores indicating accepting behavior for item 31 and rejecting behavior for item 32; items 33-34 1=Extremely to 5=Not At All with higher scores indicating accepting behavior for item 33 and rejecting behavior for item 34.
  LGBTQ Microaggressions and Microaffirmations in Families - interpersonal negative (microaggression) subscale is 8 items with a 5 point scale 0=Never to 4=All the time. Higher scores suggest experiencing more interpersonal microaggressions.
(Intermediary Outcome) Outness (Youth) | No time frame at pre-test (enrollment), post-test (within one week of intervention end), or 6-month follow-up.
  Nebraska Outness Scale- Differentiating disclosure and concealment in measurement of outness for sexual minorities is a 12 item measure with 2 subscales of 6 items each (sexual orientation and gender identity). 11 point scale 0=0% to100=100%. Higher scores indicate greater disclosure of outness.
(Intermediary Outcome) Internalized homo/bi/trans phobia (Youth) | No time frame at pre-test (enrollment), post-test (within one week of intervention end), or 6-month follow-up.
  Items from the 2017 LGBTQ+ Teen Survey includes 4 items on a 4 point scale 1=Strongly disagree to 4=Strongly agree. Higher scores indicate increased feelings of internalized homo/bi/trans phobia.
(Intermediary Outcome) Hope for the future (Youth) | No time frame at pre-test (enrollment), post-test (within one week of intervention end), or 6-month follow-up.
  Items from the 2017 LGBTQ+ Teen Survey Hope for the future is a 4 item measure with a 4 point scale 1=Definitely no to 4=Definitely yes. Higher scores indicate higher levels of hope and optimism.
(Intermediary Outcome) Parent-child prevention related conversations (Youth and Caregivers) | No time frame at pre-test (enrollment), post-test (within one week of intervention end), or 6-month follow-up.
  Items adapted from Edwards et al. (2022) is an 11 item measure with a 4 point scale 1=Strongly disagree to 4=Strongly agree. Higher scores indicate more frequent healthy parent/child prevention related/focused conversations.
(Intermediary Outcome) Positive ethnic/racial identity (Youth and Caregivers) | No time frame at pre-test (enrollment), post-test (within one week of intervention end), or 6-month follow-up.
  Multi-group Ethnic Identity Scale is a 12 item measure on a 4 point scale 1=Strongly disagree to 4=Strongly agree. Higher scores indicate increased positive feelings of racial and ethnic identity.
(Intermediary Outcome) Positive LGBTQ+ Identity (Youth) | No time frame at pre-test (enrollment), post-test (within one week of intervention end), or 6-month follow-up.
  Lesbian, Gay, and Bisexual Positive Identity Measure is a 5 item measure on a 7 point scale 1=Strongly disagree to 7=Strongly agree. Higher scores indicate stronger sense of LGBTQ+ identity and social justice.
(Intermediary Outcome) Caregiver of LGBTQ+ Youth Positive Identity (Caregivers) | No time frame at pre-test (enrollment), post-test (within one week of intervention end), or 6-month follow-up.
  adapted Lesbian, Gay, and Bisexual Positive Identity Measure is a 5 item measure on a 7 point scale 1=Strongly disagree to 7=Strongly agree. Higher scores indicate stronger sense of their youth's LGBTQ+ identity and social justice.
(Intermediary Outcome) Caregiver - Youth Communication (Youth and Caregivers) | No time frame at pre-test (enrollment), post-test (within one week of intervention end), or 6-month follow-up.
  Parent-Adolescent Communication Scale is a 20 item measure with a 5 point scale 1=Strongly disagree to 5=Strongly agree. Higher scores indicate more positive adolescent-parent communication.
(Intermediary Outcome) Sense of Community (Youth and Caregivers) | No time frame at pre-test (enrollment), post-test (within one week of intervention end), or 6-month follow-up.
  Sense of Community Index 2 (SCI-2) is a 25 item measure. Item 1 has a 6 point scale 1= I'd prefer not to be part of this community -- 6= Very important to me. 24 items have a 4 point scale 0=Not at all -- 3=Completely. Higher scores indicate a sense of belonging and purpose in the LGBTQ community.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No